CLINICAL TRIAL: NCT03987685
Title: A Dose Regimen-Finding Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Activity of Oral Topotecan With HM30181A Monotherapy in Patients With Advanced Malignancies
Brief Title: Evaluate Oral Topotecan With HM30181A Monotherapy in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORATOP-001
Record Dates: First submitted 2019-01-08; First posted 2019-06-17 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2019-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oratopo (Experimental): To determine the Maximum Tolerated Dose (MTD) of oral topotecan with HM30181A administered once daily for 5 consecutive days every 21 days.
  Interventions: Drug: Oratopo

INTERVENTIONS:
Drug: Oratopo — Oral topotecan will be supplied in topotecan capsules and oral HM30181A-US tablets
  Other Names: oral topotecan + oral HM30181A

SUMMARY:
This is a multicenter, nonrandomized, open-label, safety, tolerability and pharmacokinetic (PK) study to determine the MTD and optimal dosing of Oratopo. No control group has been included.

DETAILED DESCRIPTION:
This is a multicenter, open-label, safety, tolerability, pharmacokinetic, and activity study. Eligible subjects will be adults with advanced solid tumor malignancies. In the treatment period groups of 3 to 6 subjects will receive a single dose of oral Oratopo will be administered and will be followed for toxicity. Dose escalation will continue until an MTD is reached, or nonlinear increases in exposure are confirmed, or a maximum dose of Oratopo is reached.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male and female adults ≥18 years of age
* Histologically or cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Topotecan monotherapy is a reasonable treatment in the judgement of the Investigator
* Measurable disease as per RECIST v1.1 criteria
* Able to swallow oral medication as an intact dosage form
* Adequate hematologic status as demonstrated by not requiring transfusion support or granulocyte colony-stimulating factor (G-CSF)levels maintained
* Adequate liver function.
* Adequate renal function
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Life expectancy of at least 3 months
* Females must be postmenopausal (>12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or, if sexually active, must be using effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 30 days after their last dose of study drug.
* Sexually active male patients must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 30 days after the last dose of study drug.

Exclusion Criteria:

* Currently taking a prohibited concomitant medication, other than a premedication, that are Strong inhibitors or strong inducers of cytochrome P450
* Unresolved toxicity from prior chemotherapy
* Planning to receive other medical, surgical, or radiological cancer treatments during the course of this study
* Received investigational agents within 14 days or 5 half-lives prior to the first study dosing day, whichever is longer
* Require therapeutic use of anticoagulants.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, clinically significant myocardial infarction unstable angina pectoris, clinically significant cardiac arrhythmia, bleeding disorder, chronic pulmonary disease requiring oxygen, or psychiatric illness/social situations that would limit compliance with study requirements.
* Major surgery to the upper GI tract
* Hypersensitivity to topotecan or allergy to HM30181A or its excipients.
* Any other condition which the Investigator believes would make participation in the study not acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2021-01-09 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) | Day 1 through 21
  dose limiting toxicities occuring in the first cycle of therapy

SECONDARY OUTCOMES:
Safety assessment using Adverse Events of Oratopo | Weekly, from randomization throughout the study for approximately 24 months
  Safety assessment using Adverse Events of Oratopo
Pharmacokinetics of Oratopo | At the end of Cycle 1 (each cycle is 21 days)
  Plasma concentrations of Oratopo

CONTACTS AND LOCATIONS:
Overall Officials: David Cutler, MD, Study Director — Athenex, Inc.
Locations (3):
- HonorHealth Research Institute, Phoenix, Arizona, United States
- United Kingdom (2):
  - Cancer Research UK Clinical Trials Unit- The Beatson West of Scotland Cancer Centre, Glasgow
  - Sir Bobby Robson Cancer Trials Research Centre, Freeman Hospital, Newcastle

IPD SHARING:
Plan to Share IPD: No